CLINICAL TRIAL: NCT02257970
Title: Placebo-controlled, Case-controlled, Open Label Therapeutic Trial for Unilateral or Bilateral Lymphedema of Arm or Leg.
Brief Title: Lymphedema Study for Arm or Leg Lymphedema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine; Professor of Cardiovascular Medicine, Stanford University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7781
Record Dates: First submitted 2014-08-25; First posted 2014-10-07 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Lymphedema
Keywords: Lymphedema; edema; swelling
MeSH Terms: conditions — Lymphedema; Edema | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1: Exploratory Group (Experimental): Ketoprofen 225-300 mgs daily, taken orally
  Ketoprofen-exploratory group: 225-300 mgs daily for four to six months
  Interventions: Drug: Ketoprofen
- Part 2: Open-label Group (Experimental): Ketoprofen 225 mg daily, taken orally
  Open-label group: 75 mgs, three times daily, for four months
  Interventions: Drug: Ketoprofen
- Part 3: Placebo Group (Placebo Comparator): Participants randomized to receive placebo: placebo, three times daily, taken orally
  Placebo: 1 capsule, three times daily, for four months
  Interventions: Drug: Placebo
- Part 3: Ketoprofen Group (Active Comparator): Participants randomized to receive active medication: ketoprofen 75 mgs., three times daily, taken orally
  Ketoprofen: 1 capsule, three times daily, for four months
  Interventions: Drug: Ketoprofen

INTERVENTIONS:
Drug: Ketoprofen
  Arms: Part 1: Exploratory Group; Part 2: Open-label Group; Part 3: Ketoprofen Group
Drug: Placebo — Placebo to match ketoprofen.
  Arms: Part 3: Placebo Group

SUMMARY:
This study compares the effectiveness of a study drug versus placebo in the treatment of lymphedema.

DETAILED DESCRIPTION:
Part 1 is feasibility, exploratory, open-label study of ketoprofen, to document effects.

Part 2, is open-label trial of ketoprofen to document histological response. Part 3 is double-blind randomized trial of receive placebo or ketoprofen to evaluate safety and efficacy.

We will try to determine how the study drug affects the body tissue by obtaining tissue biopsies (small pieces of skin from the arm or leg) before treatment and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* a history of lymphedema of one or more limbs (unilateral or bilateral), with a duration of > 6 months.

Exclusion Criteria:

* Patients with active cancer, infection or bleeding tendency will be excluded.
* We will also exclude patients with medical contraindications to NSAIDs, including history of allergies, know gastrointestinal intolerance, or other serious systemic illness (e.g., renal failure, hepatic dysfunction, congestive heart failure, neurological or psychological impairment) that would impair the patients' ability to participate.
* Minors (<18 years of age) *>90 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-03; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Rockson SG, Tian W, Jiang X, Kuznetsova T, Haddad F, Zampell J, Mehrara B, Sampson JP, Roche L, Kim J, Nicolls MR. Pilot studies demonstrate the potential benefits of antiinflammatory therapy in human lymphedema. JCI Insight. 2018 Oct 18;3(20):e123775. doi: 10.1172/jci.insight.123775. PMID 30333315
- See also: Stanford Health Care: Center for Lymphatic and Venous Disorders — http://stanfordhealthcare.org/medical-clinics/center-lymphatic-venous-disorders.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 was feasibility, exploratory, open-label ketoprofen, to document effects. Part 2 was open-label trial of ketoprofen to document histological response. Part 3 was double-blind randomized to receive placebo or ketoprofen to evaluate safety and efficacy.
Period: Part 1
Arm/Group | Part 1: Exploratory Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
Started | 50 | 0 | 0 | 0
Completed | 50 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Exploratory Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
Started | 0 | 23 | 0 | 0
Completed | 0 | 16 | 0 | 0
Not Completed | 0 | 7 | 0 | 0
Period: Part 3
Arm/Group | Part 1: Exploratory Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
Started | 0 | 0 | 23 | 21
Completed | 0 | 0 | 16 | 14
Not Completed | 0 | 0 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Participants that completed the protocol were included in Baseline Characteristics.
Groups:
- Part 2: Open-label Group: Ketoprofen 225 mg daily
  Open-label group: 75 mgs, 1 capsule, taken orally, three times daily, for four months
- Part 3: Placebo Group: Participants randomized to receive placebo:
  1 capsule, taken orally, three times daily, for four months
- Part 3: Ketoprofen Group: Participants randomized to receive active medication, Ketoprofen 225 mg daily:
  Ketoprofen: 75 mgs, 1 capsule, three times daily, for four months
- Total: Total of all reporting groups
Arm/Group | Part 1: Exploratory Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group | Total
Number analyzed (Participants) | 50 | 16 | 16 | 14 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 12 | 14 | 10 | 75
  >=65 years | 11 | 4 | 2 | 4 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.72 (13.46) | 56.43 (11.15) | 50.25 (15.12) | 53.92 (13.14) | 54.92 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 13 | 14 | 14 | 82
  Male | 9 | 3 | 2 | 0 | 14
Lymphedema classification [Count of Participants; unit: Participants] — Primary lymphedema is defined as having been born with the condition, or developed the condition in the first year of life.
  Secondary lymphedema is defined as a condition that results due to some other event (e.g., trauma, cancer treatment, May-Turner Syndrome (MTS)).
  Participants
    Primary | 4 | 5 | 4 | 2 | 15
    Secondary | 46 | 11 | 12 | 12 | 81
Lymphedema location [Count of Participants; unit: Participants]
  Upper extermity | 18 | 4 | 5 | 2 | 29
  Lower extremity | 32 | 12 | 11 | 12 | 67

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Count of Participants Able to Complete Ketoprofen Treatment
Description: Participants who were able to complete ketoprofen treatment and experienced no treatment-related serious adverse events.
Time Frame: Baseline to month 6
Population: This outcome was assessed in Part 1 participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Exploratory Group
Number analyzed (Participants) | 50
Participants | 50

2. Primary Outcome: Part 2: Change From Baseline in Cutaneous Histological Architecture
Description: Quantitative assessment of paired histological specimens of lymphedema skin pre- and post-treatment with ketoprofen. The impact of treatment on cutaneous histopathology was evaluated through the use of an empirically-derived scoring system (comprised of dermal thickness, intercellular mucin content, deep dermal collagen content, and perivascular infiltrate); this quantitative assessment was developed and performed by a dermatopathologist. Each characteristic was weighted equally and each specimen was assigned a cumulative subscale score of 0-5. The scores were summed for a total score (range: 0-20) which is presented here. Higher scores indicate a higher degree of pathology. A quantitatively higher negative change indicates a more favorable therapeutic response in the histology.
Time Frame: Baseline; Month 4
Population: This primary endpoint outcome was assessed in Part 2 participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 2: Unaffected Tissue Samples: Results from normal samples from Part 2 participants are presented in this reporting group.
Arm/Group | Part 2: Open-label Group | Part 2: Unaffected Tissue Samples
Number analyzed (Participants) | 16 | 16
score on a scale
  Baseline | 6.125 (2.247) | 0.8 (1.2)
  Month 4 | 2.688 (1.401) | 0.6 (1.0)
Statistical Analysis 1: Comparison: Part 2: Open-label Group; For the analysis, the 4-month post-minus-pre change in this score for ketoprofen was compared; Test type: Equivalence — The likelihood of rejecting the null hypothesis (equivalence between the two groups) was defined as P<0.05; p < 0.0001, t-test, 2 sided; paired t-test

3. Primary Outcome: Part 3: Measurement of Skin Thickness
Description: Caliper-measured skin thickness (mm) was serially assessed and pre-to-post paired analysis was performed for both arms (Placebo and Ketoprofen) of the study.
Time Frame: Baseline and 4 months
Population: Data for this outcome were collected in Part 3 participants only and for lymphedema-affected limbs only.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
Number analyzed (Participants) | 16 | 14
mm
  Baseline | 47 (28) | 49 (21)
  Month 4 | 45 (31) | 41 (21)
Statistical Analysis 1: Comparison: Part 3: Placebo Group; Test type: Equivalence — Pre-to-post comparison: the likelihood of rejecting the null hypothesis (equivalence between the two groups) was defined as P<0.05; p = 0.6, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Part 3: Ketoprofen Group; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.01, t-test, 2 sided; paired t-test

4. Secondary Outcome: Part 2: Measurement of Skin Thickness
Description: Caliper measured skin thickness (mm) of lymphedema-affected limb was serially assessed and pre-to-post paired analysis was performed.
Time Frame: Baseline and 4 months
Population: Data for this outcome were collected in Part 2 participants only and for lymphedema-affected limbs only.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 2: Open-label Group
Number analyzed (Participants) | 16
mm
  Baseline | 62 (34)
  Month 4 | 27 (22)

5. Secondary Outcome: Part 3: Change From Baseline in Cutaneous Histological Architecture
Description: Quantitative assessment of paired histological specimens of lymphedema skin pre- and post-treatment with ketoprofen or placebo, respectively. The impact of treatment on cutaneous histopathology was evaluated through the use of an empirically-derived scoring system (comprised of dermal thickness, intercellular mucin content, deep dermal collagen content, and perivascular infiltrate); this quantitative assessment was developed and performed by a dermatopathologist. Each characteristic was weighted equally and each specimen was assigned a cumulative subscale score of 0-5. The scores were summed for a total score (range: 0-20) which is presented here. Higher scores indicate a higher degree of pathology. For the analysis, the 4-month post-minus-pre change in this score for ketoprofen- and placebo-recipients, respectively, was compared. A quantitatively higher negative change indicates a more favorable therapeutic response in the histology.
Time Frame: Baseline; 4 months
Population: Data for this outcome were collected in Part 3 participants only and for lymphedema tissue samples only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 3 Placebo: Placebo, 1 capsule taken orally, three times daily, for four months
- Part 3: Ketoprofen Group: Ketoprofen, 75 mgs, 1 capsule taken orally, three times daily, for four months
- Part 3: Unaffected Tissue Samples: Results from normal samples from Part 3 participants are presented in this reporting group.
Arm/Group | Part 3 Placebo | Part 3: Ketoprofen Group | Part 3: Unaffected Tissue Samples
Number analyzed (Participants) | 16 | 14 | 30
score on a scale
  Baseline | 2.7 (2.1) | 4.1 (1.8) | 0.8 (1.2)
  Month 4 | 1.0 (1.1) | 1.18 (1.08) | 0.6 (1.0)

6. Secondary Outcome: Part 2/Part 3: Change From Baseline in Bioimpedance Spectroscopy
Description: A four-electrode configuration was used to non-invasively assess the extracellular and intracellular fluid contents of the limb. Data were analyzed according to Cole theory, using the manufacturer's software (Impedimed Ltd.), to provide values for a bioimpedance ratio (Ro), the resistance of the extracellular fluid including lymph, R∞ the resistance of total tissue fluid and Ri, the resistance of the intracellular fluid. For the purposes of these investigations, in patients with unilateral lymphedema, the ratio of Ro in the affected:unaffected limbs was analyzed in each patient, as a measure of the bioimpedance attributable to the extracellular fluid content. An Ro level of 1.034 was considered normal; values ≥1.034 were considered abnormal.
Time Frame: Baseline; 4 months
Population: Data for this outcome were collected for Part 2 and Part 3 participants with unilateral lymphedema-affected limbs only.
Measure: Mean (Standard Deviation); unit: ratio of Ro values
Units Other Than Participants: limbs
Groups:
- Part 3: Placebo Group: Participants randomized to receive placebo:
  1 capsule, three times daily, for four months
- Part 3: Ketoprofen Group: Participants randomized to receive active medication:
  Ketoprofen 75 mgs., 1 capsule, taken orally, three times daily, for four months
Arm/Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
Number analyzed (Participants) | 10 | 12 | 13
Number analyzed (limbs) | 20 | 24 | 26
ratio of Ro values
  Baseline | 1.5 (0.5) | 1.5 (0.4) | 1.4 (0.2)
  Month 4 | 1.6 (0.3) | 1.5 (0.3) | 1.4 (0.2)

7. Secondary Outcome: Part 2/Part 3: Change in Limb Volume
Description: Quantitative assessment of limb volume (ml) of the affected limb at study end compared to pre-treatment values.
Time Frame: Baseline; 4 months
Population: Data for this outcome were collected only for lymphedema-affected limbs only.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
Number analyzed (Participants) | 16 | 16 | 14
ml
  Baseline | 9866 (5821) | 7196 (3519) | 8598 (3066)
  Month 4 | 9465 (5115) | 7256 (3496) | 8675 (3103)

8. Secondary Outcome: Part 3: Change in Systemic Inflammatory Mediator Granulocyte Colony Stimulating Factor (G-CSF)
Description: The systemic inflammatory response of G-CSF, in the two treatment groups, Ketoprofen and Placebo, will be assessed with Luminex-bead inflammasome analysis of pre- and post-treatment plasma samples. G-CSF, a glycoprotein, is an inflammatory cytokine produced by endothelium and immune cells. Ketoprofen is a unique NSAID possessing dual pathways of inflammatory inhibition, blocking cyclooxygenase (COX) and 5-LO. Measurement using median fluorescence intensity (MFI) was employed.
Time Frame: Baseline; 4 months
Population: Data for this outcome was collected for Part 3 participants only.
Measure: Mean (Standard Deviation); unit: MFI (log10)
Groups:
- Part 3: Placebo: Placebo, 1 capsule taken orally, three times daily, for four months
Arm/Group | Part 3: Placebo | Part 3: Ketoprofen Group
Number analyzed (Participants) | 16 | 14
MFI (log10)
  Baseline | 121 (90) | 131 (76)
  Month 4 | 209 (214) | 126 (107)

ADVERSE EVENTS:
Time Frame: Four months
Arm/Group | Part 1: Exploratory Group | Part 2: Open-label Group | Part 3: Placebo Group | Part 3: Ketoprofen Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/23 | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/23 | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 3/50 | 2/23 | 1/23 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1: Exploratory Group (N=50) | Part 2: Open-label Group (N=23) | Part 3: Placebo Group (N=23) | Part 3: Ketoprofen Group (N=21)
Cellulitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1/19 (1)
Hemorrhoidal hemorrhag (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No